CLINICAL TRIAL: NCT03381833
Title: A Multi-Center, Randomized, Open-Label, Parallel-Group Study With LJPC-401 for the Treatment of Myocardial Iron Overload in Patients With Transfusion-Dependent Beta Thalassemia
Brief Title: A Study With LJPC-401 for the Treatment of Myocardial Iron Overload in Patients With Transfusion-Dependent Beta Thalassemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated early for lack of efficacy as determined by interim endpoint analyses
Sponsor: La Jolla Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LJ401-BT01
Record Dates: First submitted 2017-12-12; First posted 2017-12-22 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Beta-Thalassemia
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A - Delayed therapy (Active Comparator): standard chelation therapy alone for 26 weeks followed by standard chelation therapy plus LJPC-401 for 26 weeks
  Interventions: Drug: LJPC-401
- Group B - Immediate therapy (Active Comparator): standard chelation therapy plus LJPC-401 for 52 weeks
  Interventions: Drug: LJPC-401

INTERVENTIONS:
Drug: LJPC-401 — subcutaneous injection, up to 20 mg per week from week 26 to 52
  Other Names: synthetic human hepcidin
  Arms: Group A - Delayed therapy
Drug: LJPC-401 — subcutaneous injection, up to 20 mg per week from week 1 to 52
  Other Names: synthetic human hepcidin
  Arms: Group B - Immediate therapy

SUMMARY:
This study is a Phase 2 multicenter, randomized, open-label, parallel-group study. The primary objective of the study is to evaluate the effect of LJPC-401 (synthetic human hepcidin) on iron levels in patients with transfusion-dependent beta thalassemia with myocardial iron overload.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 14 years of age with transfusion-dependent beta thalassemia.
* Patients must have increased iron levels in the heart as measured by magnetic resonance imaging (MRI). Two separate cardiac T2*MRI from 6 to 35 msec; <= 15% difference between the two.
* Patients must be receiving iron chelation therapy for a minimum of 1 year and be on a stable dose prior to study and expected to remain stable during study.
* Female patients of childbearing potential must not be pregnant, must have negative pregnancy tests, and must use an effective birth control method during the study.
* Male patients must be either surgically sterile or use an effective birth control method during the study.
* Patient must be willing and able to provide written informed consent. Parent of legal guardian to patients younger than age of majority must be willing and able to provide informed consent.

Exclusion Criteria:

* Any significant medical condition or lab abnormality that would prevent the patient from participating in the study.
* Pregnant or lactating women.
* Patients taking an immunosuppressive agent (except topical over-the-counter steroids, inhaled steroid medications, and non-steroidal anti-inflammatory drugs) or have a planned surgery (except dental surgery or simple dermatologic procedures).
* Patients participating in an unapproved investigational clinical trial within 30 days of this study.
* Patients with a disease, disability or condition which may interfere with the conduct of the study, or which would, in the opinion of the Investigator, pose an unacceptable risk to the patient.
* Patients who are unwilling or unable to comply with the study requirements.
* Patients with known hepatitis B or hepatitis C, or being treated for a positive viral load or are noncompliant with hepatitis medications.
* Known and active human immunodeficiency virus (HIV) infection.
* Patients with Child Pugh class C cirrhosis or liver failure.
* Patients with severe congestive heart failure (NYHA Class 4).
* Use of erythropoiesis stimulating agents in the past 3 months prior to study entry.
* History of allergic reaction to hepcidin or excipients.
* Contraindication to MRI scanning.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2020-01-14 (Actual)

PRIMARY OUTCOMES:
Effect of LJPC-401 on cardiac iron | 26 Weeks
  Change in cardiac T2* magnetic resonance imaging (MRI)

SECONDARY OUTCOMES:
Effect of LJPC-401 on cardiac iron | 52 Weeks
  Change in cardiac T2*MRI
Effect of LJPC-401 on hepatic iron | 52 Weeks
  Change in hepatic T2*MRI
Effect of LJPC-401 on serum iron | 56 Weeks
  Mean change in serum iron
Effect of LJPC-401 on hemoglobin | 52 Weeks
  Mean change in hemoglobin
Effect of LJPC-401 on volume of blood transfused | 56 Weeks
  Change in transfused blood volume
Effect of LJPC-401 on its potential to elicit an immune response | 56 Weeks
  Measured by blood laboratory tests and the presence of anti-drug antibodies
Effect of LJPC-401 on the incidence of treatment-emergent adverse events | 56 Weeks
Effect of LJPC-401 on vital signs-heart rate | 56 Weeks
Effect of LJPC-401 on vital signs-body temperature | 56 Weeks
Effect of LJPC-401 on vital signs-respiratory rate | 56 Weeks
Effect of LJPC-401 on vital signs-blood pressure | 56 Weeks
Effect of LJPC-401 on body weight | 56 Weeks
  Change in body weight (kilograms)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (2):
  - Investigative Site, Oakland, California
  - Investigative Site, New York, New York
- Australia (2):
  - Investigative Site, Camperdown, New South Wales
  - Investigative Site, Liverpool, New South Wales
- Greece (3):
  - Investigative Site, Goudi, Attica
  - Investigative Site, Thessaloniki, Macedonia
  - Investigative Site, Patra, Peloponnese
- Italy (5):
  - Investigative Site, Cagliari
  - Investigative Site, Modena
  - Investigative Site, Napoli
  - Investigative Site, Orbassano
  - Investigative Site, Verona
- Investigative Site, Beirut, Lebanon
- Thailand (2):
  - Investigative Site, Bangkok Noi
  - Investigative Site, Chiang Mai
- Turkey (Türkiye) (4):
  - Investigative Site, Adana
  - Investigative Site, Ankara
  - Investigative Site, Antalya
  - Investigative Site, Izmir
- United Kingdom (2):
  - Investigative Site, London, England
  - Investigative Site, London

IPD SHARING:
Plan to Share IPD: No